CLINICAL TRIAL: NCT05871099
Title: Hyperthermic Intraperitoneal Chemotherapy in the Treatment of Locally Advanced Gastric Cancer After Laparoscopic Gastrectomy With D2 Lymphadenectomy: A Phase III Multicenter Prospective Randomized Controlled Clinical Trial
Brief Title: Laparoscopic Gastrectomy With D2 Lymphadenectomy Combined With Hyperthermic Intraperitoneal Chemotherapy (HIPEC) or Not
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Collaborators: Shandong Cancer Hospital and Institute (Other); Chinese PLA General Hospital (Other); Zibo Central Hospital (Other Government); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Jinan Central Hospital (Other); Qilu Hospital of Shandong University (Other); Yantai Yuhuangding Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Shandong First Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); Hebei Medical University Fourth Hospital (Other); Peking University Cancer Hospital & Institute (Other); Peking University People's Hospital (Other); Tianjin Cancer Hospital (Unknown); First Affiliated Hospital Xi'an Jiaotong University (Other); Union Hospital of Huazhong University of Science and Technology (Unknown); Wuhan University (Other); Brigham and Women's Hospital (Other); Second Xiangya Hospital of Central South University (Other); Weihai Municipal Hospital (Other); Mountain University Cancer Hospital (Unknown); Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIPEC-09
Record Dates: First submitted 2023-05-14; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Gastric Cancer
Keywords: Advanced Gastric Cancer; HIPEC; Laparoscopic Gastrectomy; Randomized Clinical Trial; Recurrence-free survival
MeSH Terms: conditions — Stomach Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group receive laparoscopic (robotic) D2 surgery plus HIPEC2 times plus systemic chemotherapy 6~8 cycles.
  Interventions: Procedure: Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
- Control group (No Intervention): Control group receive laparoscopic (robotic) D2 surgery + systemic chemotherapy 6-8 cycles

INTERVENTIONS:
Procedure: Hyperthermic Intraperitoneal Chemotherapy (HIPEC) — Experimental group receive HIPEC two times after laproscopic gastrectomy
  Arms: Experimental group

SUMMARY:
The goal of this clinical trial is to learn about Hyperthermic Intraperitoneal Chemotherapy in the Treatment of Locally Advanced Gastric Cancer after Laparoscopic Gastrectomy with D2 Lymphadenectomy. The main question it aims to answer is: whether HIPEC can effectively improving the 5-year overall survival rate and decrease the peritoneal metastases rate of patients with advanced gastric cancer underwent Laparoscopic Gastrectomy with D2 Lymphadenectomy. Participants will be divided into two groups, Experimental group received laparoscopic (robotic) D2 surgery plus HIPEC2 times plus systemic chemotherapy 6~8 cycles; and Control group received laparoscopic (robotic) D2 surgery plus systemic chemotherapy 6~8 cycles.

ELIGIBILITY:
Inclusion Criteria:

(1) Newly treated patients who did not receive chemotherapy, radiotherapy or other antitumor therapy before the start of the clinical trial;(2) Aged 18-80 years;(3) male or non-pregnant or lactating female;(4) Gastric adenocarcinoma was pathologically confirmed, and laparoscopic (robotic) radical gastrectomy was planned;(5) Patients with T stage T3 or above, no distant metastasis, and feasible criteria for laparoscopic D2 radical resection (AJCC Eighth edition);(6) The estimated survival time is more than 6 months;(7) History of nonabdominal surgery (except laparoscopic cholecystectomy);(8) The bone marrow reserve function was good, and the blood routine met the following conditions: white blood cell count ≥3.5×109/L, neutrophil ≥1.5×109/L, platelet count ≥100×109/L, hemoglobin ≥90g/L;(9) Organ function was good, and biochemical examination met the following conditions: ALT≤2.5× upper limit of normal value (ULN), AST≤2.5×ULN, serum total bilirubin ≤1.5×ULN, serum creatinine ≤1.5×ULN;(10) Functional status: 0-1 (ECOG);(11) Preoperative ASA grade I-III;(12) Voluntarily sign the informed consent.

Exclusion Criteria:

(1) Lymph node BulkyN2 status was diagnosed by abdominal CT/MRI, that is, at least one lymph node meridian ≥3cm or three consecutive lymph nodes, each meridian ≥1.5cm;(2) pregnant or lactating women;(3) Other malignant tumors within 5 years;(4) Preoperative temperature ≥38℃ or complicated with infectious diseases requiring systematic treatment;(5) serious mental illness;(6) Severe respiratory diseases, FEV1< 50%;(7) Severe liver and kidney dysfunction, liver enzyme elevation more than 2 times the normal value;(8) History of unstable angina pectoris or myocardial infarction within 6 months;(9) History of cerebral infarction or cerebral hemorrhage within 6 months, except old infarct;(10) Systemic glucocorticoid therapy within 1 month;(11) Patients with gastric cancer complications (bleeding, perforation, obstruction) requiring emergency surgery;(12) The patient has participated in or is currently participating in other clinical studies (within 6 months);(13) Laparoscopic exploration, biopsy and cytology confirmed intraperitoneal implantation and metastasis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Estimated)
Dates: Start 2022-11-20 (Actual); Primary Completion 2024-11-20 (Estimated); Study Completion 2039-11-20 (Estimated)

PRIMARY OUTCOMES:
5-years Recurrence-free survival | 5 years

SECONDARY OUTCOMES:
5-year overall survival rate | 5 years
peritoneal metastasis rate | 5 years
peritoneal metastasis-free survival | 5 years
Regional recurrence rate | 5 years
  local recurrence after radical gastrectomy refers to the recurrence of anastomosis, duodenal stump, tumor bed, and residual stomach, including the recurrence of regional lymph nodes
distant metastasis rate | 5 years
Toxic and side effects of the program | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yanbing Zhou, MD, Study Director — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR